CLINICAL TRIAL: NCT00644995
Title: Step Up Wellness Program for Depression, Physical Inactivity, and Smoking
Brief Title: Effectiveness of The Step Up Wellness Program for People With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH080658 (NIH); R34MH080658 (NIH)
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: Depression; Smoking; Physical Activity
MeSH Terms: conditions — Depression; Smoking; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Control (Active Comparator): Participants will receive usual care which includes advice to stop smoking and referral to standard care treatment available through participants' health insurance and health plan.
  Interventions: Behavioral: Usual care
- Step Up Intervention (Experimental): Participants will receive the Step Up Wellness Program. The intervention is detailed below.
  Interventions: Behavioral: Step Up Wellness Program

INTERVENTIONS:
Behavioral: Step Up Wellness Program — Participants in the Step Up Wellness program will receive weekly phone calls from a study health coach. During these calls, the coach will discuss ways to improve and manage mood, increase physical activity, and prepare to quit smoking.
  Arms: Step Up Intervention
Behavioral: Usual care — Participants will receive referral usual care treatment for depression and smoking cessation, plus self-help physical activity intervention.
  Arms: Usual Care Control

SUMMARY:
This randomized pilot study will evaluate the feasibility and acceptability of a phone-based wellness program for improving mood, physical activity, and smoking abstinence rates among people with depression who also are physically inactive and smoke cigarettes.

DETAILED DESCRIPTION:
This pilot study will evaluate the feasibility, acceptability, and potential effectiveness of the Step Up Wellness Program among people with depression who also are physically inactive and smoke cigarettes.

Participation in this study will last 6 months. All participants will complete a baseline survey and then be assigned randomly to receive the Step Up Wellness Program or usual care for 3 months. Participants in the Step Up program will receive weekly phone calls from a study health coach. During these calls, the coach will discuss ways to improve and manage mood, increase physical activity, and prepare to quit smoking. Participants will also be given materials to review and homework assignments between calls. Participants in the usual care group will receive standard care which includes referrals for treatment of depression and nicotine dependence, as well as self-help information on physical activity. All participants will be surveyed at 4 and 6 months post-enrollment. Participants will also provide qualitative feedback on the program.

ELIGIBILITY:
Inclusion Criteria:

* Member of Group Health insurance plan
* Aged 18 to 75
* Experiencing at least moderate depressive symptoms
* Low physical activity defined as failure to meet Centers for Disease Control (CDC) guidelines for weekly activity OR low to moderate physical activity as assessed by International Physical Activity Questionnaire (IPAQ)
* Current smoker
* Has a phone
* Able to read and speak in English
* No mobility or physical impairments that would prevent engaging in moderate physical activity
* Without a hearing impairment that would prevent participation with the phone-based counseling or assessments

Exclusion Criteria:

* Self-report of bipolar disorder or schizophrenia
* Currently receiving specialty mental health care or smoking cessation treatment
* If on an antidepressant, has been taking it less than 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McClure, PhD, Principal Investigator — Group Heatlh Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Result] McClure JB, Catz SL, Ludman EJ, Richards J, Riggs K, Grothaus L. Feasibility and acceptability of a multiple risk factor intervention: the Step Up randomized pilot trial. BMC Public Health. 2011 Mar 17;11:167. doi: 10.1186/1471-2458-11-167. PMID 21414216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Group Health, a large regional health plan.Potential participants were identified from automated medical records, mailed study invitation letters, and then contacted by phone to be screened for interest and eligibility.
Groups:
- Usual Care: Advice to quit and referral to standard care
- Step Up: proactive phone counseling addressing smoking, depression, and PA
Period: Overall Study
Arm/Group | Usual Care | Step Up
Started | 25 | 27
Completed 4 Month Assessment | 23 | 24
Completed | 23 (Completed 6 month assessment) | 23
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 4
Not completed — Refused | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Advice to quit smoking and referral to standard care
- Step Up: Proactive phone counseling addressing smoking, depression, and physical activity (PA)
- Total: Total of all reporting groups
Arm/Group | Usual Care | Step Up | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (11.8) | 43.5 (11.8) | 44.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Depression Score
Description: % with significant change (50% reduction in SCL [Symptom Checklist] depression score)
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- Step Up: Proactive phone counseling addressing smoking, depression and physical activity
Arm/Group | Usual Care | Step Up
Number analyzed (Participants) | 23 | 24
percentage of participants | 13 [lower limit 1.85] | 52

2. Primary Outcome: Abstinent From Smoking
Description: self-reported 7 day point prevalent abstinence with non-responders coded as smokers
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- Step Up: Proactive phone counseling addressing smoking, depression and PA
Arm/Group | Usual Care | Step Up
Number analyzed (Participants) | 25 | 27
percentage of participants | 20 | 11

3. Primary Outcome: Days Walk Per Week
Description: Mean change in days walk per week from baseline
Time Frame: 6 months
Measure: Mean (Full Range); unit: mean change in days walked per week
Arm/Group | Usual Care | Step Up
Number analyzed (Participants) | 23 | 23
mean change in days walked per week | 0.74 [-4.0 to 7.0] | 1.13 [-5.0 to 7.0]

4. Primary Outcome: Minutes Per Week of Moderate Physical Activity
Description: Mean change from baseline as assessed using International Physical Activity Questionnaire (IPAQ)
Time Frame: 6 months
Measure: Mean (Full Range); unit: mean change in minutes per week of PA
Arm/Group | Usual Care | Step Up
Number analyzed (Participants) | 23 | 23
mean change in minutes per week of PA | 96 [-360 to 1500] | 121 [-600 to 2520]

5. Primary Outcome: Minutes Per Week of Vigorous Physical Activity
Description: Mean change from baseline assessed using IPAQ physical activity scale
Time Frame: 6 months
Measure: Mean (Full Range); unit: minutes per week
Arm/Group | Usual Care | Step Up
Number analyzed (Participants) | 23 | 23
minutes per week | 60 [-45.0 to 360.0] | 3 [-960.0 to 480.0]

6. Secondary Outcome: Number of Cigarettes Smoked Per Day
Description: Mean change in cigarettes smoked per day from baseline
Time Frame: 4 months
Measure: Mean (Full Range); unit: mean change in number of cigs/day smoked
Arm/Group | Usual Care | Step Up
Number analyzed (Participants) | 25 | 27
mean change in number of cigs/day smoked | -1.8 [-14.0 to 10.0] | -3.2 [-20.0 to 5.0]

7. Secondary Outcome: Quit Attempt
Description: % who made a quit attempt, defined as intentionally not smoking for at least 24 hours
Time Frame: 6 months
Measure: Number; unit: percent of participants
Arm/Group | Usual Care | Step Up
Number analyzed (Participants) | 23 | 23
percent of participants | 65 | 83

ADVERSE EVENTS:
Groups:
- Step Up: Proactive phone counseling addressing smoking, depression, and physical activity
Arm/Group | Usual Care | Step Up
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

LIMITATIONS AND CAVEATS:
This was a pilot feasibility trial and was not powered to detect statistically significant outcomes.

Point prevalent abstinence outcomes imputed missing values as smokers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes